CLINICAL TRIAL: NCT01539031
Title: Randomized, Multicenter, Double-blind, Double-dummy, Parallel-Group Study With an Open-label Extension Phase to Compare the Efficacy and Safety of Donepezil Hydrochloride 23 mg Treatment With Continuation of Donepezil Hydrochloride 10 mg Treatment in Japanese Subjects With Severe Alzheimer's Disease
Brief Title: Compare the Efficacy and Safety of Donepezil Hydrochloride 23 mg Treatment With Continuation of Donepezil Hydrochloride 10 mg Treatment in Japanese Subjects With Severe Alzheimer's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: E2020-J081-343
Record Dates: First submitted 2012-02-21; First posted 2012-02-27 (Estimated); Last update posted 2023-06-18 (Actual); Status verified 2015-09

CONDITIONS: Alzheimer's Type Dementia
Keywords: Alzheimer Disease; Dementia; Delirium; Amnestic; Cognitive Disorders; Donepezil; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Tauopathies; Neurodegenerative Diseases; Mental Disorders; Cholinesterase Inhibitors; Enzy
MeSH Terms: conditions — Alzheimer Disease; Dementia; Delirium; Cognitive Dysfunction; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Tauopathies; Neurodegenerative Diseases; Mental Disorders | interventions — Donepezil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 10 mg group (Experimental)
  Interventions: Drug: E2020
- 23 mg group (Active Comparator)
  Interventions: Drug: E2020

INTERVENTIONS:
Drug: E2020 — Subjects in the Group-10 mg:
  Week 1 to 4: Once daily donepezil 10 mg and placebo matching donepezil 5 mg, Week 5 to 28: Once daily donepezil 10 mg and placebo matching donepezil 23 mg, Week 29 to 32: Once daily donepezil 5 mg, 10 mg and placebo matching donepezil 23 mg, Week 33 to 52: Once daily donepezil 23 mg
  Arms: 10 mg group
Drug: E2020 — Subjects in the Group-23 mg:
  Week 1 to 4: Once daily donepezil 5 mg and 10 mg, Week 5 to 28: Once daily donepezil 23 mg and placebo matching donepezil 10 mg, Week 29 to 32: Once daily donepezil 23 mg, and placebo matching donepezil 5 mg and 10 mg, Week 33 to 52: Once daily donepezil 23 mg
  Arms: 23 mg group

SUMMARY:
The purpose of this study is to compare 23 mg donepezil sustained release to the currently marketed formulation of 10 mg donepezil immediate release in patients with severe Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria

* Diagnosis: diagnostic evidence of probable Alzheimer's disease (AD) consistent with Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV-TR) 290.00 or 290.10
* Mini Mental State Examination (MMSE) less than or equal to 12 and greater than or equal to1 inclusive, at Screening
* SIB less than or equal to 90 and greater than or equal to10 at both Screening and Baseline
* No evidence of focal disease to account for dementia on any cranial image (magnetic resonance imaging [MRI] or computed tomography [CT]).
* Subject age range: male and female subjects greater than or equal to 50 years of age inclusive
* Outpatients (patients in nursing homes are eligible)
* The subject must have a caregiver who will provide informed consent separately for his/her own participation in the study, who will have regular contact with the subject.
* Stable donepezil dose of 10 mg, taken as a single, daily dose for greater than or equal to 3 months prior to the Screening visit
* Subjects who can swallow hole tablets, as tablets should not be broken or crushed
* Comorbid medical conditions must be clinically stable prior to Screening unless otherwise specified.
* Written informed consent will be obtained from the subject (if possible) or from the subject's legal guardian or other representative (according to Japanese regulations as appropriate) prior to beginning screening activities.

Exclusion Criteria

* Subjects with a known history of disorders that affect cognition or the ability to assess cognition but are distinguishable from AD
* Subjects with dementia complicated by other organic disease or AD with delirium
* Known hypersensitivity to donepezil or piperidine derivatives, or to any of the excipients in the study drug formulation
* Patients who are expected to live in a nursing home within 24 weeks after randomization (eligible if temporary)
* Use of any prohibited prior or concomitant medications. Memantine will be allowed if taken at prescribed doses that are less than or equal to 20 mg/day, provided that the dose has been stable for at least 6 months prior to Screening.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 351 (Actual)
Dates: Start 2012-03; Primary Completion 2015-01 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
The Severe Impairment Battery (SIB) | 24 weeks
  SIB: change from Baseline to Week 24 in the total SIB score - Last Observation Carried Forward (LOCF)
The Clinician's Interview-Based Impression of Change, Plus Caregiver Input Version (CIBIC+) | 24 weeks
  CIBIC+: overall change score at Week 24 - Last Observation Carried Forward (LOCF)

CONTACTS AND LOCATIONS:
Overall Officials: Naoki Kubota, Study Director — Neuroscience Clinical Development Section, Japan/Asia Clinical Research Product Creation Unit, Eisai Product Creation Systems, Eisai Co., Ltd.
Locations (54):
- Japan (54):
  - Anjo, Aichi-ken
  - Ōbu, Aichi-ken
  - Toyoake, Aichi-ken
  - Chikushi, Fukuoka
  - Kitakyushu, Fukuoka
  - Fukuoka, Gunma
  - Miyoshi, Hiroshima
  - Ōtake, Hiroshima
  - Amagasaki, Hyōgo
  - Himeji, Hyōgo
  - Morioka, Iwate
  - Numakunai, Iwate
  - Kida, Kagawa-ken
  - Takamatsu, Kagawa-ken
  - Kawasaki, Kanagawa
  - Sagamihara, Kanagawa
  - Yokohama, Kanagawa
  - Yokosuka, Kanagawa
  - Maizuru, Kyoto
  - Nagasaki, Kyushu
  - Sendai, Miyagi
  - Kitamorokata, Miyazaki
  - Ina, Nagano
  - Nagaoka, Niigata
  - Kurashiki, Okayama-ken
  - Ibaraki, Osaka
  - Ikeda, Osaka
  - Sakai, Osaka
  - Sennan, Osaka
  - Takatsuki, Osaka
  - Age, Saitama
  - Iruma, Saitama
  - Kasukabe, Saitama
  - Tokorozawa, Saitama
  - Fuji, Shizuoka
  - Izunokuni, Shizuoka
  - Anan, Tokushima
  - Bunkyo-ku, Tokyo
  - Kodaira, Tokyo
  - Koto, Tokyo
  - Ōta-ku, Tokyo
  - Setagaya City, Tokyo
  - Suginami, Tokyo
  - Akita
  - Chiba
  - Fukuoka
  - Hiroshima
  - Kagoshima
  - Kochi
  - Kyoto
  - Nara
  - Osaka
  - Saitama
  - Tokushima